CLINICAL TRIAL: NCT03785743
Title: Total Laparoscopic Pancreaticoduodenectomy Versus Open Pancreaticoduodenectomy for Pancreatic Carcinoma(TJDBPS07) a Multicenter Randomized Controlled Trial
Brief Title: Comparing Laparoscopic and Open Surgery for Pancreatic Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Shandong Provincial Hospital (Other Government); The Second Hospital of Hebei Medical University (Other); The Affiliated Hospital of Xuzhou Medical University (Other); Xinqiao Hospital of Chongqing (Other); Hunan Provincial People's Hospital (Other); The First Hospital of Jilin University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); The Third Affiliated Hospital of Soochow University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Afﬁliated Hospital of North Sichuan Medical College (Other); First Affiliated Hospital of Chongqing Medical University (Other); Peking Union Medical College Hospital (Other); Henan Provincial People's Hospital (Other); Sir Run Run Shaw Hospital (Other); Fujian Medical University Union Hospital (Other); Fudan University (Other)
Responsible Party: Principal Investigator, Renyi Qin, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJDBPS07
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Pancreatic Carcinoma; Laparoscopic; Pancreaticoduodenectomy
Keywords: Pancreatic Carcinoma; Laparoscopic; Pancreaticoduodenectomy; Survival
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLPD (Experimental): Total laparoscopic pancreaticoduodenectomy for pancreatic cancer
  Interventions: Procedure: TLPD Surgery
- OPD (Experimental): Open pancreaticoduodenectomy for pancreatic cancer
  Interventions: Procedure: OPD Surgery

INTERVENTIONS:
Procedure: TLPD Surgery — TLPD
  Arms: TLPD
Procedure: OPD Surgery — OPD
  Arms: OPD

SUMMARY:
Background: Pancreatic cancer (PC) is one of the most aggressive malignant neoplasms with poor outcomes. Pancreatoduodenectomy (PD) is the only curative treatment for PC. Minimally invasive surgery has been progressively developed, first with the advent of hybrid-laparoscopy and recently with the total laparoscopy surgeries, but a number of issues are currently being debated, including the superiority between total laparoscopic pancreaticoduodenectomy (TLPD)and the open pancreaticoduodenectomy (OPD). Studies comparing these two surgery techniques are merging and randomized controlled trials (RCT) are lacking but clearly required.

Methods/design: TJDBPS07 is a multicenter prospective, randomized controlled, trial comparing TLPD and OPD in pancreatic cancers. A total of 200 patients with pancreatic cancer underwent PD will be randomly allocated to the TLPD group or OPD group with an enhanced recovery after surgery (ERAS) pattern. The trial's aim is to exploring the overall survival (OS), disease free survival (DFS) and quality of life. The duration of the entire trial is seven years including prearrangement, a presumably five-year follow-up and analyses.

Discussion: Despite the fact there are several RCTs comparing minimally invasive pancreaticoduodenectomy (MIPD) and Open approach or LPD versus OPD. This trial will be the first comparing TLPD and OPD in a large multicenter setting. TJDBPS01 trial is hypothesized to assess whether TLPD has superiority over OPD in recovery and other aspects.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 years and 75 years.
2. Histologically confirmed PDAC or clinically diagnosed PDAC by an MDT without histopathologic evidence.
3. Patients feasible to undergo both LPD and OPD according to MDT evaluations.
4. Patients understanding and willing to comply with this trial.
5. Provision of written informed consent before patient registration.
6. Patients meeting the curative treatment intent in accordance with clinical guidelines.

Exclusion Criteria:

1. Patients with distant metastases, including peritoneal, liver, distant lymph node metastases, and involvement of other organs.
2. Patients requiring left, central or total pancreatectomy or other palliative surgery.
3. Preoperative American Society of Anaesthesiologists (ASA) score ≥ 4.
4. History of other malignant disease.
5. Pregnant or breast-feeding women.
6. Patients with serious mental disorders.
7. Patients treated with neoadjuvant therapy.
8. Patients with vascular invasion and requiring vascular resection as evaluated by the MDT team according to abdominal imaging data.
9. Body mass index > 35 kg/m2.
10. Patients participating in any other clinical trials within 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 year
  5-year overall survival

SECONDARY OUTCOMES:
overall survival | 5 years
  the interval between the day of surgery and the day of death for various reasons
disease-free survival | 5 years
  the interval between the day of surgery and the day of tumour recurrence
90-day mortality | 90 days
  the percentage of patients who died within 90 days postoperatively
complication rate | 90 days
  complications related to PD
comprehensive complication index | 90 days
  calculated as the sum of all complications that are weighted for their severity
length of stay | 90 days
  the number of nights spent in the hospital from the end of the surgical procedure until discharge or death
intraoperative indicators | 90 days
  description of the patients' intraoperative condition relating to the safety of patients

CONTACTS AND LOCATIONS:
Overall Officials: Renyi Qin, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Biliary and Pancreatic Surgery, Tongji Hospital, Affiliated Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang M, Pan S, Qin T, Xu X, Huang X, Liu J, Chen X, Zhao W, Li J, Liu C, Li D, Liu J, Liu Y, Zhou B, Zhu F, Ji S, Cheng H, Li Z, Li J, Tang Y, Peng X, Yu G, Chen W, Ma H, Xiong Y, Meng L, Lu P, Zhang Z, Yu X, Zhang H, Qin R. Short-Term Outcomes Following Laparoscopic vs Open Pancreaticoduodenectomy in Patients With Pancreatic Ductal Adenocarcinoma: A Randomized Clinical Trial. JAMA Surg. 2023 Dec 1;158(12):1245-1253. doi: 10.1001/jamasurg.2023.5210. PMID 37878305
- [Derived] Pan S, Qin T, Yin T, Yu X, Li J, Liu J, Zhao W, Chen X, Li D, Liu J, Li J, Liu Y, Zhu F, Wang M, Zhang H, Qin R; Minimally Invasive Treatment Group in the Pancreatic Disease Branch of China's International Exchange and Promotion Association for Medicine and Healthcare (MITG-P-CPAM). Laparoscopic versus open pancreaticoduodenectomy for pancreatic ductal adenocarcinoma: study protocol for a multicentre randomised controlled trial. BMJ Open. 2022 Apr 4;12(4):e057128. doi: 10.1136/bmjopen-2021-057128. PMID 35379633